CLINICAL TRIAL: NCT05120739
Title: Skin Preparation of Patients Before Orthopedic Surgery : A Randomized Controlled Study on the Efficacy of Chlorhexidine Cloths Versus Chlorhexidine Soaps
Brief Title: Efficacy of CHX Cloths Versus CHX Soaps for Bathes Before Orthopedic Surgery
Acronym: POL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 38RC19.254
Record Dates: First submitted 2021-10-26; First posted 2021-11-15 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Orthopedic Surgery
Keywords: chlorhexidine; cloths; orthopedic surgery; preoperative bath

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Skin preparations (the day before and the morning of the operation) with the 2% CHX cloths
  Interventions: Drug: 2% CHX cloths
- Control (No Intervention): Skin preparations (the day before and the morning of the operation) with the 4% CHX soap (standard of care)

INTERVENTIONS:
Drug: 2% CHX cloths — skin preparation in 2% CHX cloths
  Arms: Interventional

SUMMARY:
Surgical site infections (SSI) in orthopedic surgery are rare events but associated with great morbidity as well as a significant additional cost. The World Health Organization (WHO) recently carried out meta-analyzes on all the existing prophylactic measures and could not rule on the use of chlorhexidine (CHX) cloths due to the low number of studies available. CHX cloths could actually benefit patients for whom preoperative showering is not possible, whether in emergency or trauma settings due to pain-induced functional impotence. A randomized controlled clinical study aimed at evaluating the in vivo microbiological efficacy of CHX cloths in a population of orthopedic surgery patients while evaluating the psycho-social determinants of adherence to a new preoperative preparation technique seems essential.

ELIGIBILITY:
Inclusion Criteria:

* adult patients,
* undergoing orthopedic surgery: programmed hip prosthesis (non-urgent),
* admitted the day before the operation
* and having given their written consent.

Exclusion Criteria:

* presence of a documented infection at the time of the intervention,
* presence of skin wounds,
* presence of antibiotic treatment within 15 days before the operation
* intolerance to CHX,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Relative decrease in the number of bacterial colonies before the antiseptic preparation of the operating site at the surgical room (T1) | Between the patient's admission to the CHU GA and just before the antiseptic preparation of the operating site at the surgical room (Day 1)
  Relative decrease in the number of bacterial colonies measured between the patient's admission to the Grenoble Alps University Hospital (CHU GA) (T0) and after 2 preoperative skin preparations (the day before and the morning of the operation), and just before the antiseptic preparation of the operating site at the surgical room (T1) in the 2% CHX cloths group versus the 4% CHX soap group.

SECONDARY OUTCOMES:
Relative decrease in the number of bacterial colonies after 1 preoperative skin preparation | Between the patient's admission to the CHU GA and after 1 preoperative skin preparation (Day 0)
  Relative decrease in the number of bacterial colonies measured between the patient's admission to the CHU GA (T0) and after 1 preoperative skin preparation (the day before the evening of the operation)
Relative decrease in the number of bacterial colonies after 2 preoperative skin preparations | Between the patient's admission to the CHU GA and after 2 preoperative skin preparations (Day 1)
  Relative decrease in the number of bacterial colonies measured between the patient's admission to the CHU GA (T0) and after 2 preoperative skin preparations (the night before and the morning of the operation)
Significant predictors of a decrease in bacterial colonization | Between the patient's admission to the CHU GA and just before the antiseptic preparation of the operating site at the surgical room (Day 1)
  Significant predictors of a decrease in bacterial colonization among the sex, age of the patients, their co-morbidities, the use of cloths and the time between the last preoperative skin preparation and the skin sample in the operating room
Percentage of skin adverse reactions | Between the patient's admission to the CHU GA and just before the antiseptic preparation of the operating site at the surgical room (Day 1)
  Percentage of skin adverse reactions after 2 preoperative skin preparations in the 2% CHX cloths group versus the 4% CHX soap group.
Nursing load | Between the patient's admission to the CHU GA and just before the antiseptic preparation of the operating site at the surgical room (Day 1)
  Nursing load in the 2% CHX cloths group versus 4% CHX soap group according to the Soins Infirmiers Individualisés à la Personne Soignée (SIIPS) scale
Duration of preoperative skin preparation | Between the patient's admission to the CHU GA and just before the antiseptic preparation of the operating site at the surgical room (Day 1)
  Duration of preoperative skin preparation in minutes in the 2% CHX cloths group versus 4% CHX soap group.
Responses to a questionnaire for patients and adherence score | Between surgery and discharge from the hospital (Day 4)
  Responses to a questionnaire for patients and adherence score in the 2% CHX cloths group versus the 4% CHX soap group.
Responses to a semi-structured interview intended for healthcare professionals | Interview at the end of the inclusion of patients (through study completion, an average of 6 months)
  Responses to a semi-structured interview intended for healthcare professionals who cared for patients randomized to the 2% CHX cloths group versus the 4% CHX soap group.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Grenoble Alpes, Grenoble, France

REFERENCES:
- [Derived] Gallouche M, Rubens-Duval B, Boisset S, Margotton M, Caspar Y, Le Marechal M, Bosson JL, Astagneau P, Gauchet A, Landelle C. Evaluation of microbiological efficacy of 2% chlorhexidine gluconate cloths versus 4% chlorhexidine gluconate soap for preoperative preparation/shower in total joint arthroplasty: a single-centre randomised controlled trial. Antimicrob Resist Infect Control. 2025 Nov 25;14(1):143. doi: 10.1186/s13756-025-01661-z. PMID 41291848